CLINICAL TRIAL: NCT06774378
Title: Efficacy of an Occupational Intervention for Quality of Work Life in ADHD: A Randomized Controlled Trial Protocol
Brief Title: Efficacy of an Occupational Intervention for Improving Quality of Work Life in Adults Living With ADHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Collaborators: Fonds de recherche du Québec - Société et culture (Unknown)
Responsible Party: Principal Investigator, Geneviève Sauvé, Assistant Professor, Université du Québec a Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-0SYA-312580
Record Dates: First submitted 2024-11-26; First posted 2025-01-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: ADHD
Keywords: ADHD; RCT; intervention; quality of life; work; mental health; workplace; quality of work life
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Minds@Work-ADHD-Quality of Life
  Interventions: Behavioral: Minds@Work-ADHD-Quality of Life
- Control (Placebo Comparator): Minimal contact comparison approach
  Interventions: Behavioral: Minimal contact

INTERVENTIONS:
Behavioral: Minds@Work-ADHD-Quality of Life — Minds@Work-ADHD-Quality of Life
  Arms: Intervention
Behavioral: Minimal contact — Weekly 15-minute scripted phone calls made individually by a member of the research team to offer minimal support, without any active intervention.
  Arms: Control

SUMMARY:
An adaptation of the Minds@Work intervention to improve quality of life at work for adults living with attention deficit disorder with/without hyperactivity (ADHD), following a group format.

DETAILED DESCRIPTION:
In this study, the research team has developed a psychosocial group intervention specifically aimed at improving quality of life at work for ADHD workers. Work-related themes cover motivation, accommodations, problem solving, cognitive functions (i.e. attention and memory), hyperactivity and impulsivity, interpersonal interactions, and medication management.

The general objective of this project is to evaluate the effectiveness of this new psychosocial intervention aimed at improving the quality of life at work of workers living with ADHD, using a randomized controlled trial design.

More specifically, the project will aim to:

Objective #1: Evaluate the effectiveness of the intervention on the quality of life at work of workers living with ADHD (primary outcome).

Objective #2: Evaluate the effectiveness of the intervention on secondary variables, namely the satisfaction of psychological needs, job satisfaction, well-being at work, self-esteem as a worker, occupational self-efficacy, cognitive functioning, self-compassion and the quality of the relationship with members of the workplace (secondary outcomes).

* Hypothesis #1: There will be a statistically significant improvement in the quality of life at work between the pre- and post-intervention measurements in participants receiving the experimental condition.
* Hypothesis #2: There will be a statistically significant condition*time interaction indicating that the improvement in quality of work life among participants receiving the experimental condition between the pre- and post-intervention measurement times will be greater than that of the control condition.
* Hypotheses #3 to 10: There will be a statistically significant improvement in the secondary outcomes mentioned above between the pre- and post-intervention measurements among participants receiving the experimental condition.
* Hypothesis #11: For participants receiving the experimental condition, there will be no statistically significant difference in quality of work life between the follow-up times, indicating that the gains acquired during the intervention will be maintained at 3, 6, 9, and 12 months.

Our research team collaborates with the PANDA Les Deux-Rives association, which is a non-profit organization specializing in ADHD. The psychosocial intervention was co-designed, which allows the involvement of field stakeholders in all stages of the research. This involvement promotes the creation of a final research output that will meet the needs of the target population and that will be easily implemented in the organizational structures already in place.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* French language proficiency
* Score ≤ 4 on Part A of the Adult ADHD Self-Report Scale (ASRS-v1.1)
* Currently employed
* Express desire to improve Quality of Work Life (QoWL)

Exclusion Criteria:

* Currently receiving psychosocial services (e.g., psychotherapy, occupational therapy) specifically targeting QoWL improvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Work Life as Measured by Quality of Work Life Questionnaire (QWLQ) Total Score | Assessed at baseline (pre-intervention), immediately after the intervention, and at 3, 6, 9, and 12 months post-intervention
  The QWLQ will be used to assess multiple dimensions of work-related quality of life, including work tasks, workplace environment and conditions, self-esteem as a worker, sense of belonging to a workgroup, and relationships with coworkers/supervisors. The questionnaire consists of 40 items rated on a 4-point Likert scale (1 = completely disagree to 5 = completely agree). Total scores range 40-200, with higher scores indicating greater perceived quality of work life.

SECONDARY OUTCOMES:
Change in Psychological Need States at Work Scale (PNSW-S) Score | Assessed at baseline (pre-intervention), immediately after the intervention, and at 3, 6, 9, and 12 months post-intervention
  The PNSW-S assesses satisfaction, frustration, and unfulfillment of basic psychological needs (autonomy, competence, relatedness) in the workplace. The 37-item questionnaire uses a Likert scale, with higher scores (Min = 37, Max = 259) indicating greater psychological need satisfaction. The scale measures intrinsic motivation based on self-determination theory.
Change in Minnesota Satisfaction Questionnaire-Short Form (MSQ-SF) Scores | Assessed at baseline (pre-intervention), immediately after the intervention, and at 3, 6, 9, and 12 months post-intervention
  The MSQ-SF is a 20-item measure assessing three domains: Intrinsic Job Satisfaction (task-related attitudes), Extrinsic Job Satisfaction (working conditions/environment), and General Satisfaction. Items are rated on a Likert scale, with higher scores indicating greater job satisfaction in each domain (Min = 20, Max = 100) .
Change in Index of Psychological Well-Being at Work (IPWBW) Score | Assessed at baseline (pre-intervention), immediately after the intervention, and at 3, 6, 9, and 12 months post-intervention
  The IPWBW is a 25-item measure assessing five dimensions of well-being at work: Interpersonal Fit, Thriving, Feeling of Competency, Desire for Involvement, and Perceived Recognition at Work. Items are rated on a Likert scale, with higher scores indicating greater psychological well-being at work (Min = 0, Max = 100) .
Change in Individual Self-Esteem as a Worker (ISEW) Scale Score | Assessed at baseline (pre-intervention), immediately after the intervention, and at 3, 6, 9, and 12 months post-intervention
  The ISEW is a 10-item scale measuring individual and social dimensions of worker self-esteem. Items are rated on a Likert scale, with higher scores indicating greater self-esteem as a worker (Min = 10, Max = 40).
Change in Occupational Self-Efficacy Scale-Short Version (OSES) Score | Assessed at baseline (pre-intervention), immediately after the intervention, and at 3, 6, 9, and 12 months post-intervention
  The OSES is a 6-item measure assessing workers' sense of self-efficacy based on Bandura's self-efficacy theory. Items are rated on a Likert scale, with higher scores indicating greater occupational self-efficacy (Min = 6, Max = 36).
Change in Self-Compassion Scale-Short Form (SCS-S) Score | Assessed at baseline (pre-intervention), immediately after the intervention, and at 3, 6, 9, and 12 months post-intervention
  The SCS-S is a 12-item measure assessing self-kindness, self-judgment, and feelings of loneliness. Items are rated on a Likert scale, with higher scores indicating greater self-compassion in work settings (Min = 12, Max = 60).
Change in Cognitive Function at Work Questionnaire (CFWQ) Score | Assessed at baseline (pre-intervention), immediately after the intervention, and at 3, 6, 9, and 12 months post-intervention
  The CFWQ is a 29-item measure assessing subjective cognitive difficulties in six domains: Memory, Language, Executive Function, Speed of Processing, Cognitive Control, and Name Memory. Items are rated on a Likert scale, with higher scores indicating better cognitive functioning at work (Min = 0, Max = 58).
Change in Team-Member Exchange (TMX) Survey Score | Assessed at baseline (pre-intervention), immediately after the intervention, and at 3, 6, 9, and 12 months post-intervention
  The TMX is a 9-item survey measuring the quality of professional relationships between adults with ADHD and workplace stakeholders. Items are rated on a Likert scale, with higher scores indicating better quality of work relationships (Min = 9, Max = 63).

OTHER OUTCOMES:
Professional Situation Assessment: Job Tenure and Strategy Implementation | Assessed at 3, 6, 9, and 12 months after completing the 8-week intervention
  A follow-up survey assessing two components: (1) job tenure status and (2) implementation of workplace strategies. Control group participants complete 2 items and intervention group participants complete 3 items to characterize their professional situation. Responses will track job retention and use of learned strategies in the workplace.

CONTACTS AND LOCATIONS:
Locations (1):
- Université du Québec à Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
For this project, IPD sharing is not included in the ethical approval provided by our Institutional Review Board (IRB).

REFERENCES:
- [Background] Sauve G, Buck G, Lepage M, Corbiere M. Minds@Work: A New Manualized Intervention to Improve Job Tenure in Psychosis Based on Scoping Review and Logic Model. J Occup Rehabil. 2022 Sep;32(3):515-528. doi: 10.1007/s10926-021-09995-2. Epub 2021 Jul 30. PMID 34331191
- [Derived] Voyer C, Corbiere M, Villotti P, Stamate AN, Sauve G. Efficacy of an occupational intervention for quality of work life in ADHD: A randomized controlled trial protocol. Contemp Clin Trials. 2025 Aug;155:107997. doi: 10.1016/j.cct.2025.107997. Epub 2025 Jun 30. PMID 40602661